CLINICAL TRIAL: NCT04587427
Title: Drug utilisatIon Study of Radium 223 Under Routine Clinical Practice in Europe
Brief Title: A Study to Learn More About How Radium-223 is Being Used With Other Treatments in European Patients Who Have Not Received Radium-223 Before
Acronym: DIRECT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20702
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Bone Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223: Subjects who received the treatment of radium-223 during the before or after label change study periods.
  Interventions: Drug: Radium 223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium 223 dichloride (Xofigo, BAY88-8223) — Prescribed by physicians.

SUMMARY:
In this study data from people with metastatic castration-resistant prostate cancer (mCRPC) with bone metastasis are studied. mCRPC is a prostate cancer which has spread to other parts of the body even when the amount of testosterone in the body was reduced. Bone metastasis is when the cancer has spread to the bones.

The study drug, radium-223, is currently available as a treatment for mCRPC with bone metastasis. But, its combination with certain other cancer treatments may lead to medical problems. Therefore the instructions about how doctors should use radium-223 with other cancer treatments were changed.

In this study, the researchers want to learn more about how doctors are now using radium-223 to treat patients with mCRPC and bone metastasis.

The participants in this study will include men in Denmark, Germany, or the Netherlands. They will not have received radium-223 before. They will have at least 6 months of medical records before starting treatment with radium-223. The researchers will collect the participants' medical records up to December 2020.

The researchers will review information from the participants' medical records and medical claims from hospitals where the participants received radium-223. They will look at the medical records of participants who first started receiving radium-223 before there were new instructions about using it with other cancer treatments. They will also look at the medical records of participants who first started receiving radium-223 after there were new instructions.

They will then count how many participants received other specific cancer treatments with radium-223. They will compare the results of the participants' who received radium-223 before the new instructions and those who received it after the new instructions.

There are no required visits or tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive a first dispensing/administration of radium-223 during the before or after study period
* Patients who have at least 6 months of continuous enrolment in the study databases before the first dispensing/administration of radium-223 (to allow for evaluation of recent medical history and medication use)

Exclusion Criteria:

* Patients who used radium-223 ever before the start of the before study period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include new users of radium-223 during the study periods captured in each data source. The study period will include time periods before and after the label change. The "before" period will start in November 2013, the month of radium-223 approval, and will end the in November 2017, the month when the first Direct Healthcare Professional Communication (DHCP) letter was sent. The "after" period will include an enrolment phase during which patients initiating radium-223 in each data source will be identified. The enrolment phase will last at least 1 year, starting in April 2019 (6 months after the label change), and will continue through a follow up phase of at least 6 months after the last new user of radium-223 is identified.
Sampling Method: Non-Probability Sample
Enrollment: 1067 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who use radium-223 in combination with abiraterone acetate | Data will be collected from Nov 2013 to Dec 2020
The proportion of patients who use radium-223 in combination with other systemic therapies for mCRPC, except luteinising hormone-releasing hormone (LHRH) analogues | Data will be collected from Nov 2013 to Dec 2020
The proportion of patients who use radium-223 without having received at least two prior lines of systemic therapy for mCRPC, except LHRH analogues | Data will be collected from Nov 2013 to Dec 2020

SECONDARY OUTCOMES:
The difference between before and after the label change periods in the proportion of patients who use radium-223 in combination with abiraterone acetate | Data will be collected from Nov 2013 to Dec 2020
The difference between before and after the label change periods in the proportion of patients who use radium-223 in combination with other systemic therapies for mCRPC, except luteinising hormone-releasing hormone (LHRH) analogues | Data will be collected from Nov 2013 to Dec 2020
The difference between before and after the label change periods in the proportion of patients who use radium-223 without having received at least two prior lines of systemic therapy for mCRPC, except LHRH analogues | Data will be collected from Nov 2013 to Dec 2020

OTHER OUTCOMES:
Descriptive summary of patient characteristics | Data will be collected from Nov 2013 to Dec 2020
  Including:
  * Age (in years)
  * Calendar year when radium-223 was first prescribed/dispensed, as recorded in each data source
  * Time since first available prostate cancer diagnosis
  * Confirmed diagnosis (yes/no) of mCRPC
  * Prior use (yes/no) systemic therapy for CRPC
  * Prior use (yes/no) systemic therapy for hormone-sensitive prostate cancer (HSPC)
  * Presence of metastasis at baseline: bone or visceral
  * Total level of serum alkaline phosphatase, when available: as U/L and categorised as above or below a threshold (e.g., < 220 U/L and ≥ 220
  U/L):
  * Prior use of bone-health agents (yes/no) since first diagnosis of PC
  * Prior use of systemic corticosteroids: yes/no, since first diagnosis of PC
  * History (diagnosis or treated for osteoporosis) of osteoporosis ever before the index date

CONTACTS AND LOCATIONS:
Locations (3):
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Netherlands

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.